CLINICAL TRIAL: NCT02711293
Title: The Impact of Home Delivery of Antiretroviral Therapy on Virological Suppression: A Non-inferiority Cluster-randomized Controlled Trial in Dar es Salaam, Tanzania
Brief Title: The Impact of Home Delivery of Antiretroviral Therapy on Virological Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Management and Development for Health (Unknown); International Initiative for Impact Evaluation (Other)
Responsible Party: Principal Investigator, Till Barnighausen, Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RIDIE-STUDY-ID-562a718b12fa0
Record Dates: First submitted 2016-03-12; First posted 2016-03-17 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: HIV; Community Health Workers; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ART home delivery + enhanced nutrition counseling (Experimental): Community health workers visit participants at home (maintaining patients' prior clinic visit frequency) to deliver antiretroviral therapy (ART) and to provide standard plus enhanced nutrition counseling.
  Interventions: Other: ART home delivery; Other: Enhanced nutrition counseling
- ART home delivery + no enhanced nutrition counseling (Experimental): Community health workers visit participants at home (maintaining patients' prior clinic visit frequency) to deliver antiretroviral therapy (ART) and to provide standard counseling.
  Interventions: Other: ART home delivery
- No ART home delivery + enhanced nutrition counseling (Experimental): Community health workers visit participants at home to provide enhanced nutrition counseling. Participants will not receive ART home delivery.
  Interventions: Other: Enhanced nutrition counseling
- Standard of care (No Intervention): Participants in this arm receive facility-based ART care and no enhanced nutrition counseling. They receive community health worker visits as per the standard of care in Dar es Salaam.

INTERVENTIONS:
Other: ART home delivery — Community health workers visit participants who are clinically stable on antiretroviral therapy (ART) at home (maintaining patients' prior clinic visit frequency) to deliver ART. Clinically stable on ART was defined as 1) taking ART for at least six months, 2) having had a CD4-cell count >350 cells/μL or a suppressed viral load at six or more months after ART initiation, and 3) the patient's most current CD4-cell count must have been >350 cells/μL or the most current viral load must have shown viral suppression, with the last measurement not taken more than 12 months ago.
  Arms: ART home delivery + enhanced nutrition counseling; ART home delivery + no enhanced nutrition counseling
Other: Enhanced nutrition counseling — Community health workers visit participants at home to provide standard counseling (focusing on family planning, prevention of HIV transmission, and ART adherence) plus enhanced nutrition counseling (covering food production and dietary advice). In addition, participants who state that they have access to a plot of land or garden to grow vegetables receive a pack of seeds (amaranth, cowpea, or pumpkin) at enrolment.
  Arms: ART home delivery + enhanced nutrition counseling; No ART home delivery + enhanced nutrition counseling

SUMMARY:
Home delivery of antiretroviral therapy (ART) by community health workers (CHWs) has the potential to reduce key barriers to ART care retention. The aim of this study is to determine whether CHW-led home delivery of ART for patients who are stable on ART combined with facility-based care for those not stable on ART is non-inferior to the standard of care (facility-based care for all ART patients) in achieving and maintaining virological suppression. The primary endpoint of this trial is the proportion of ART patients (regardless of whether they were clinically stable on ART at enrollment) who are in viral failure at the end of the study period. The non-inferiority design applies only to this primary endpoint. The margin of non-inferiority was set at a Risk Ratio (comparing intervention to control) of 1.45. This is a cluster-randomized controlled trial set in Dar es Salaam. The unit of randomization is a healthcare facility with its surrounding neighborhoods (the 'catchment area'). We matched all 48 healthcare facilities offering ART services and having affiliated public-sector CHWs in Dar es Salaam into pairs (stratified by district) based on having a similar number of patients currently on ART. In each pair, one cluster was randomized to the intervention and one to the control arm. The intervention consists of home visits by CHWs to provide counseling and deliver ART to patients who are stable on ART, while the control is the standard of care (facility-based ART care and CHW home visits at least every three months without ART home delivery). In addition, within each study arm, half of the healthcare facilities were randomized to enhanced CHW-led nutrition counseling and half to standard counseling.

ELIGIBILITY:
Inclusion Criteria:

* Having attended one of the participating healthcare facilities for ART care during the enrolment period
* Living in a neighborhood that is in the healthcare facility's catchment area

Exclusion Criteria:

* ART patients who are pregnant at the time of enrollment
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2172 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The proportion of participants in viral failure, comparing participants that received the intervention (ART home delivery if stable on ART or standard facility-based care if unstable) versus those that received the standard of care. | At the end of the study period
The mean BMI of participants in clusters assigned to standard counseling by CHWs versus those in clusters assigned to standard plus enhanced nutrition counseling. | At the end of the study period

SECONDARY OUTCOMES:
Participants' healthcare expenditures | In the last six months
Self-reported ART adherence | In the last one month
The proportion of patients with access to a plot of land who grow vegetables or fruits for their own consumption. | At the end of the study period
Diversity of dietary intake | At the end of the study period
The proportion of patients who are anemic | At the end of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Till Bärnighausen, MD ScD, Principal Investigator — Harvard School of Public Health (HSPH); Pascal Geldsetzer, MBChB MPH, Principal Investigator — Harvard School of Public Health (HSPH); Nzovu Ulenga, MD, Principal Investigator — Management and Development for Health
Locations (1):
- Management and Development for Health, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Geldsetzer P, Francis JM, Sando D, Asmus G, Lema IA, Mboggo E, Koda H, Lwezaula S, Ambikapathi R, Fawzi W, Ulenga N, Barnighausen T. Community delivery of antiretroviral drugs: A non-inferiority cluster-randomized pragmatic trial in Dar es Salaam, Tanzania. PLoS Med. 2018 Sep 19;15(9):e1002659. doi: 10.1371/journal.pmed.1002659. eCollection 2018 Sep. PMID 30231024
- [Derived] Geldsetzer P, Francis JM, Ulenga N, Sando D, Lema IA, Mboggo E, Vaikath M, Koda H, Lwezaula S, Hu J, Noor RA, Olofin I, Larson E, Fawzi W, Barnighausen T. The impact of community health worker-led home delivery of antiretroviral therapy on virological suppression: a non-inferiority cluster-randomized health systems trial in Dar es Salaam, Tanzania. BMC Health Serv Res. 2017 Feb 22;17(1):160. doi: 10.1186/s12913-017-2032-7. PMID 28228134